CLINICAL TRIAL: NCT01141998
Title: Vitamin D Substitution for Patients With Chronic Pancreatitis and Malabsorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ulrich Bang, M.D., Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bang-01
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Pancreatitis; Malabsorption Syndromes
MeSH Terms: conditions — Pancreatitis, Chronic; Malabsorption Syndromes | interventions — Calcium, Dietary; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Calcium, Dietary; Radiation: UV-filtered light.; Drug: Cholecalciferol
- Vitamin D administered orally (Active Comparator)
  Interventions: Drug: Calcium, Dietary; Drug: Cholecalciferol; Radiation: UV-filtered light.
- Vitamin D administered via UVB (Experimental)
  Interventions: Drug: Calcium, Dietary; Radiation: UVB; Drug: Cholecalciferol

INTERVENTIONS:
Drug: Calcium, Dietary — 400 mg calcium two times daily. From week 0 to 10 and week 14 to 52.
  Other Names: Unikalk Basic
Drug: Cholecalciferol — 38 micrograms daily. Week 0-10.
  Other Names: Unikalk Forte
  Arms: Vitamin D administered orally
Radiation: UVB — Ultraviolet radiation type B administered in a tanning bed. One time weekly.
  Other Names: Ergoline Flair 200
  Arms: Vitamin D administered via UVB
Radiation: UV-filtered light. — Light from a tanning bed but a UV-filter stops all ultraviolet radiation. One time weekly.
  Other Names: Ergoline Flair 200
  Arms: Placebo; Vitamin D administered orally
Drug: Cholecalciferol — 38 micrograms daily. From week 14 to 52.
  Other Names: Unikalk Forte

SUMMARY:
Purpose:

The overall objective of this study is to learn more about the disease chronic pancreatitis and thus contribute to better treatments. The investigators will gain this by studying the effects of vitamin D in the body immune system and bones. The investigators will also study the uptake of vitamin D through the intestine compared with the amount of vitamin D obtained through exposure to UVB rays.

The investigators have set a series of questions which the investigators want to answer with this experiment:

Do patients with chronic pancreatitis have reduced absorption of vitamin D from the gut?

* Have the two treatment methods with vitamin D, UV radiation and tablets, the same success rate?
* Does the distribution of the white blood cells change when the vitamin D level increases and does it depend on whether the patient have UVB radiation or tablet with vitamin D?
* Will patients require reduced amounts of painkillers when vitamin D level increases?
* Does vitamin D have influence on blood sugar and thus the risk of diabetes or worsening of this?
* Could vitamin D affect the blood content of inflammation markers?
* Does the patient feel better when he takes vitamin D?
* Does bone strength increase when the patients receive grants of vitamin D?

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis
* Malabsorption
* Age min. 18 y.
* 25-hydroxyvitamin D less than 75 nmol/l
* Body mass index < 30
* Consent

Exclusion Criteria:

* Acute pancreatitis
* Cirrhosis
* Ionized calcium > 1.35 mmol/l
* Heart disease
* Former resection of gastro-intestinal tract.
* Pregnancy
* Pancreatic malignant disease
* History of skin cancer
* Other than skin cancer less then 5 y prior to inclusion in study
* Chronic kidney disease
* Type I diabetes
* Hemoglobin < 5.0 mmol/l
* Participating in other studies
* Not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D | Week 0, 2, 6, 10, 14, 20, 30, 40, 52

SECONDARY OUTCOMES:
T-lymphocytes subsets. | Week 0, 10
  Subsets of T-lymphocytes including regulatory T-lymphocytes (Tregs) and CD4+ and CD8+ lymphocytes.
Ionized calcium | week 0, 2, 6, 10, 14, 20, 30, 40, 52
Parathyroid hormone | Week 0, 2, 6, 10, 14, 20, 30, 40, 52
  To evaluate bone-metabolism.
QoL score | Week 0, 10
  Evaluation of self-reported health using two questionnaires:
  QLQ-C30 QLQ-Pan(30)

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Erik B Jensen, Ph.d., Study Director — Dept. of osteoporosis, Hvidovre Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark